CLINICAL TRIAL: NCT00256243
Title: A Pilot Study of Neoadjuvant Biweekly Doxorubicin and Cyclophosphamide (AC) With GMCSF Followed by Weekly Carboplatin/Paclitaxel With Plus or Minus Trastuzumab (TC ± H) in the Treatment of Breast Cancer
Brief Title: Neoadjuvant Biweekly Treatment Followed by Weekly Treatment of Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rita Sanghvi, Mehta (Other)
Responsible Party: Sponsor-Investigator, Rita Sanghvi, Mehta, Dr. Rita Mehta, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 03-70; 2004-3517 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Carboplatin; Granulocyte-Macrophage Colony-Stimulating Factor; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy with GM-CSF (Experimental): Doxorubicin and Cyclophosphamide (AC) Followed by Weekly Carboplatin/Paclitaxel with GM-CSF (day 2-6)
  This regimen consists of intravenous administration of doxorubicin (Adriamycin) followed by cyclophosphamide (Cytoxan) every 14 days for a total of four cycles, unless stable disease or clinical progression is documented. Two weeks after completion of the last dose of AC, weekly Carboplatin/paclitaxel will be given for 3 weeks, followed by 1 week of rest, for a total of 12. Each clinic visit will last approximately 1 hour.
  Patients who are her-2 overexpressors by FISH will also receive Trastuzumab with weekly carboplatin and paclitaxel as the combination has been found to be synergistic in advanced breast cancer with improved clinical outcome.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Carboplatin; Drug: GM-CSF; Drug: Trastuzumab

INTERVENTIONS:
Drug: Doxorubicin — 60 mg/m2 IV, bolus once every 14 days x 2-4 cycles
Drug: Cyclophosphamide — 600 mg/m2 IV once every 14 days x 2-4 cycles
Drug: Paclitaxel — 80 mg/m2 IV over 1 hour once weekly for 9-12 doses beginning two weeks after completion of last AC dose
Drug: Carboplatin — Area under the concentration curve (AUC) 2 IV once weekly for 9-12 doses beginning two weeks after completion of last AC dose
Drug: GM-CSF — 250 μg/mL IV on day 5-14 of each subcutaneous cycle of doxorubicin and injection cyclophosphamide
Drug: Trastuzumab — AUC 2 IV weekly for 12-16 doses beginning two weeks after completion of last AC dose

SUMMARY:
We proposed to use 4 cycles of AC q 2 weeks, as used in the dose dense adjuvant study with GM-CSF support on days 3-9 of the cycle. After the completion of AC we plan to administer paclitaxel and carboplatin weekly for a total of 12 doses with one week rest after every 3 weeks of treatment over 12 weeks. Patients who are her-2 over-expressors by FISH (fluorescence in situ hybridization) will also receive Trastuzumab with weekly carboplatin and paclitaxel as the combination TC±H has been found to be synergistic in advanced breast cancer with improved clinical outcome.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy, also termed primary, induction, or preoperative chemotherapy, is defined as chemotherapy administered before locoregional treatment. It was first used in locally advanced breast cancer 30 years ago. Classically, these tumors were treated with radical surgery and/or radiotherapy. However, despite this aggressive local therapy, most patients relapsed with distant metastases and eventually died (1,2). The aim of neoadjuvant therapy is to reduce the tumor volume in patients before surgical resection, thus increasing the likelihood of breast conservation. More recently, neoadjuvant therapy has been studied as a way of testing the relevance of biological markers in predicting disease outcome.

At least six randomized trials have compared survival in patients managed with either the neoadjuvant or adjuvant approaches(3,4,5,6,7,8,9). Two of the smaller trials suggested a survival advantage for patients treated with neoadjuvant chemotherapy (5,6). Other studies, including the largest trial (1523 patients) run by the NSABP, found no differences in disease-free and overall survival (4,6,9).

Induction of a pCR should be one of the primary goals of neoadjuvant therapy because patients with no evidence of tumor cells in breast and lymph nodes after treatment may have a longer disease-free and overall survival (10).

Biweekly and weekly regimens may enhance dose intensity by minimizing re-growth of cells between cycles of treatment. In fact, dose dense regimens have even shown a survival benefit in an adjuvant setting in lymph node positive breast cancer, made possible with use of G-CSF (11). There is as yet no standard best neoadjuvant treatment. Generally patients receive AC (NSABP 14) on 3-weekly regimens in neoadjuvant setting. In addition, incorporation of taxanes on a 3 weekly schedule has resulted in statistically higher pathological CR (12,13). More recently, weekly paclitaxel regimens have reported increased pathological responses compared to 3 weekly taxane regimens. Carboplatin has also emerged as an effective agent in the treatment of metastatic breast cancer (14). Moreover, the combination of carboplatin and paclitaxel has been found to be synergistic both in three-weekly regimens and weekly regimens. In fact, combination of carboplatin, paclitaxel and trastuzumab has demonstrated a survival advantage over paclitaxel and trastuzumab alone. The Phase III study, the preliminary results of which were presented at the San Antonio Breast Cancer Symposium, show that the addition of carboplatin to trastuzumab and paclitaxel resulted in a six-month improvement in the time it took for the disease to progress, compared to the standard trastuzumab and paclitaxel regimen. The study found median survival in the trastuzumab and paclitaxel arm was 33.5 months, while the group receiving the tripartite therapy had yet to reach that point after 36 months of follow-up. Furthermore, the weekly regimens of these drugs have been found to have significantly improved tolerability over three weekly regimens (15). Therefore, we propose to use 4 cycles of AC q 2 weeks, as used in the dose dense adjuvant study with GM-CSF support on days 5-14 of the cycle. After the completion of AC we plan to administer taxol and carboplatin weekly for a total of 9 doses with one week rest after every 3 weeks of treatment over 12 weeks.

Patients who are her-2 overexpressors by FISH will also receive Trastuzumab with weekly carboplatin and paclitaxel as the combination has been found to be synergistic in advanced breast cancer with improved clinical outcome.

In a separate trial, GMCSF was used in breast cancer patients treated with adriamycin based chemotherapy as the preferred growth factor in a neoadjuvant setting (16). The initial results are suggestive of improved survival of breast cancer patients given 6 versus 5 versus 4 cycles of chemotherapy with GMCSF support. Higher dendritic cell (DC) trafficking showed a trend toward improved survival. Moreover, intrapatient comparison before and after treatment showed that the percentage of S100+ DC significantly increased over the course of GM-CSF treatment. The results form the basis of current hypothesis that the primary tumor may be an in vivo antigenic stimulus for dendritic cell trafficking, and that the combination of prolonged neoadjuvant chemotherapy with GM-CSF induced immune enhancement may contribute to better tumor control and better survival.

ELIGIBILITY:
Eligibility Criteria:

1. Patients must be women with a histologically confirmed diagnosis of locally advanced or inflammatory breast carcinoma. Histologic confirmation shall be by either core needle biopsy or incisional biopsy. Punch biopsy is allowed if invasive breast cancer is documented.
2. Patients must meet one of the criteria defined below (indicate one):

   a .Selected Stage IIB (T3, N0, M0) or IIIA (T3, N1-2, M0) disease judged primarily unresectable by an experienced breast surgeon; or otherwise deemed appropriate candidates for neoadjuvant treatment.

   b. Stage IIIB (T4, Any N, M0) or (Any T, N3, M0) disease.
3. Physical examination, chest x-ray and any x-rays or scans needed for tumor assessment must be performed within 90 days prior to registration.
4. Patients with the clinical diagnosis of congestive heart failure or angina pectoris are NOT eligible. Patients with hypertension or age > 60 years must have a Multiple Gated Acquisition (MUGA) or echocardiogram scan performed within 90 days prior to registration (indicate not applicable (NA) if no MUGA required) and Left Ventricular Ejection Fraction (LVEF) % must be greater than the institutional lower limit of normal.
5. Patients must have a serum creatinine and bilirubin ≤ the institutional upper limit of normal, and an Serum glutamic oxaloacetic transaminase (SGOT) or Serum glutamic pyruvic transaminase (SGPT) ≤ 2x the institutional upper limit of normal. These tests must have been performed within 90 days prior to registration.
6. Patients must have an Absolute neutrophil count (ANC) of ≥ 1,500/μl and a platelet count of ≥ 100,000/μl. These tests must have been performed within 90 days prior to registration.
7. Patients must have a performance status of 0-2 by Zubrod criteria
8. Pregnant or nursing women may not participate due to the possibility of fetal harm or of harm to nursing infants from this treatment regimen. Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. A urine pregnancy test is required for women of childbearing potential.
9. All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-04; Primary Completion 2011-03 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mehta, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited At University of California Irvine Medical Center (UCIMC) are recruited by referral for UCIMC inpatients or outpatients.
Groups:
- Chemotherapy With GM-CSF: Doxorubicin and Cyclophosphamide (AC) Followed by Weekly Carboplatin/Paclitaxel with Granulocyte-macrophage colony-stimulating factor (GM-CSF) (day 2-6)
  This regimen consists of intravenous administration of doxorubicin (Adriamycin) followed by cyclophosphamide (Cytoxan) every 14 days for a total of four cycles, unless stable disease or clinical progression is documented. Two weeks after completion of the last dose of AC, weekly Carboplatin/paclitaxel will be given for 3 weeks, followed by 1 week of rest, for a total of 12. Each clinic visit will last approximately 1 hour.
Period: Overall Study
Arm/Group | Chemotherapy With GM-CSF
Started | 48
Completed | 38
Not Completed | 10
Not completed — Lost to Follow-up | 2
Not completed — Death | 7
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy With GM-CSF: Doxorubicin and Cyclophosphamide (AC) Followed by Weekly Carboplatin/Paclitaxel with GM-CSF (day 2-6)
  This regimen consists of intravenous administration of doxorubicin (Adriamycin) followed by cyclophosphamide (Cytoxan) every 14 days for a total of four cycles, unless stable disease or clinical progression is documented. Two weeks after completion of the last dose of AC, weekly Carboplatin/paclitaxel will be given for 3 weeks, followed by 1 week of rest, for a total of 12. Each clinic visit will last approximately 1 hour.
Arm/Group | Chemotherapy With GM-CSF
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.29 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate
Description: Clinical response (CR): Normal breast on physical exam. No mass, no thickening, no erythema, no peau d'orange.
Time Frame: 5 years
Population: Of the 48 study participants, one patient refused preoperative but received standard adjuvant AC followed by docetaxel (without trastuzumab), relapsed, and died. Therefore, 47 participants were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy With GM-CSF
Number analyzed (Participants) | 47
Participants | 47

2. Secondary Outcome: Microscopic Pathological Response Rate
Description: pathological response rate: No evidence of microscopic invasive tumor at the primary tumor site in the surgical specimen.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy With GM-CSF
Number analyzed (Participants) | 47
Participants | 47

ADVERSE EVENTS:
Time Frame: After off treatment, follow-up assessments were done every 6 months for one year. After one year, patients were followed annually for 4 more years.
Arm/Group | Chemotherapy With GM-CSF
All-Cause Mortality (participants affected / at risk) | 10/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No